CLINICAL TRIAL: NCT02166840
Title: Self Expanding Metal Stents (SEMS) or Plastic Stents to Relieve Obstruction of Obstructive Jaundice Prior to Resection of Periampullary Tumors.
Brief Title: Metal or Plastic Stents to Relieve Obstruction of Obstructive Jaundice Prior to Resection of Periampullary Tumors.
Acronym: SEMS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Lars Lundell, Professor, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2006/220-31/4; 2006/220-31/4 (Other: Regional ethics committee (EPN, Stockholm))
Record Dates: First submitted 2014-03-03; First posted 2014-06-18 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Obstructive Jaundice; Periampullary Tumour
MeSH Terms: conditions — Jaundice, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self expanding metal stent (Experimental): Patients with self expanding metal stent inserted into bile duct.
  Interventions: Procedure: Self Expanding Metal Stent
- Plastic stent (Active Comparator): Patients with obstructive jaundice who got a plastic stent inserted into bile duct.
  Interventions: Procedure: Plastic stent (7-10Fr)

INTERVENTIONS:
Procedure: Plastic stent (7-10Fr)
  Arms: Plastic stent
Procedure: Self Expanding Metal Stent
  Arms: Self expanding metal stent

SUMMARY:
Patients with obstructive jaundice due to periampullary tumor can temporarily be relieved of their jaundice with transpapillary stenting at endoscopic retrograde cholangio-pancreatography (ERCP) prior to operation. Usually plastic stents are used.

Hypothesis: Self expanding metallic stents offer a be a better alternative for preoperative stenting in patients with obstructive jaundice due to periampullary tumour obstruction.

DETAILED DESCRIPTION:
Patients who present with obstructive jaundice and have a periampullary tumor and where the patient seems to be in good condition for surgical resection are offered the opportunity to become randomized to either endoscopic drainage with self expanding metallic or plastic stents. Before randomization they are informed about the study details and have to give their consent to participate. The metallic as well as plastic stents are standard commercially available stents. Within four weeks after stent placement the patient will be operated and the following parameters will be evaluated: quality of life, clinical symptoms and lab tests. At the operation the surgeon will make an evaluation of the inflammatory reaction in the area of the bile ducts. A culture from the bile is sampled close to the area where the anastomosis will be sutured. A tissue sample is also taken from the bile ducts to evaluate inflammation. A Lymph node is also sampled for the same reason. The surgeon also evaluates the difficulty with which the stent had to be removed. Postoperative complications are monitored in line with the regular routines at the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Obstructive jaundice in periampullary tumor.

Exclusion Criteria:

* Not willing to participate.
* Not a resectable tumor.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2007-03; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Degree and amount of bile bacterial contamination at the time of resection | Time at the operation

SECONDARY OUTCOMES:
Degree of inflammation around the bile duct. | Time at the operative intervention
General complication rates | Time from intervention until day of discharge from hospital (on an average less than 90 days).
Postoperative hospital stay. | Time from intervention until day of discharge from hospital (on an average less than 90 days).
Bacterial culture of lymph nodes in the hepatoduodenal ligament. | Time of operative intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lars Lundell, Professor, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden